CLINICAL TRIAL: NCT06312579
Title: Home-based Exercise to Improve Functional Outcomes in Veterans With Recently Healed Diabetic Foot Ulcer
Brief Title: At-Home Exercise Study for Veterans With Healed Diabetic Foot Ulcers
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: E4897-P
Record Dates: First submitted 2024-02-28; First posted 2024-03-15 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Diabetic Foot Ulcer
Keywords: Clinical trial; Mobility; Diabetic foot ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This is a single center, randomized, outcome assessor blinded, parallel group clinical trial comparing a 12-week exercise regimen to standard of care.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 12-week home based exercise (Experimental): Consistent with current physical activity recommendations for older adults, participants randomized in this arm will be prescribed 5 days/week of exercise, with seated cycling exercise performed on 3 days a week (Monday, Wednesday and Friday), and strength/balance exercise performed 2 days a week (Tuesday and Thursday).
  Interventions: Behavioral: 12-week home based exercise
- 12-week standard of care (Placebo Comparator): Participants in this group will be provided with guidance on the current standard of care. This includes guidance that these patients should slowly increase ambulation with appropriately fitted footwear.
  Interventions: Behavioral: 12-week standard of care

INTERVENTIONS:
Behavioral: 12-week home based exercise — Consistent with current physical activity recommendations for older adults, participants randomized in this arm will be prescribed 5 days/week of exercise, with seated cycling exercise performed on 3 days a week (Monday, Wednesday and Friday), and strength/balance exercise performed 2 days a week (Tuesday and Thursday).
  Arms: 12-week home based exercise
Behavioral: 12-week standard of care — Participants in this group will be provided with guidance on the current standard of care. This includes guidance that these patients should slowly increase ambulation with appropriately fitted footwear.
  Arms: 12-week standard of care

SUMMARY:
Foot ulcers and amputations are a common and feared complication for people with diabetes. People with a diabetic foot ulcer have a higher risk of dying within five years than people with diabetes without an ulcer. At least one in four people with a new diabetic foot ulcer will die within five years, largely due to cardiovascular causes. The reasons for this increased mortality involve decreased mobility.

People with a recently healed diabetic foot ulcer are considered "in remission" as opposed to "cured" because the underlying medical problems which led to their ulcer are still present. Once in remission, the current standard of care is to slowly increase ambulation. The problem is that people rarely return to the recommended level of mobility. The ability to safely maintain mobility with aging is critical.

This pilot study is a small clinical trial to test the feasibility and acceptability of a home-based exercise regimen. The investigators will also assess if this home-based exercise regimen can increase mobility and function without increasing diabetic foot ulcer recurrence by improving lower extremity strength, lower extremity tissue perfusion and glycemic control.

DETAILED DESCRIPTION:
Population: 25 Veterans with a healed foot ulcer in the last 3-15 months

Site: VA Maryland Health Care System (VAMHCS)

Study Duration: Approximately 2 years

Study Design: Randomized, outcome assessor blinded, clinical trial comparing a) a 12-week home-based exercise regimen to b) standard of care

Objectives:

Primary: To assess the feasibility and acceptability of the intervention.

Secondary:

* The effect of the intervention on gait speed,
* The effect of the intervention on other measures of mobility and function including six-minute walk distance, the Modified Physical Performance Test, steps per day and community mobility, and
* The effect of the intervention on lower extremity strength, perfusion of the foot and glycemic control.

Treatment Regimens: 12-week home-based exercise regimen to standard of care

Duration of Participant's Participation: Up to 31 weeks

ELIGIBILITY:
Inclusion Criteria:

* Adults >= 50 years
* Diagnosis of diabetes
* Prior plantar foot ulcer or moderate-severe diabetic foot infection or minor lower extremity amputation.
* Two feet (can have healed minor amputations of fore and midfoot)
* Willing to wear appropriately fitted footwear for exercise regimen
* Ambulatory without walker
* Willing to enroll in the PODIMETRICS SmartMat program
* Able to give written informed consent

Exclusion Criteria:

* Unable to perform the exercise interventions (e.g. due to hearing or visual impairment)
* Anticipated foot surgery in the next 4 months
* Participating in another exercise program
* Current plantar foot ulcer or pre-ulcer
* Any other criteria which, in the investigator's opinion, would compromise the ability of a subject to participate safely

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Gait speed | 12-weeks
  Usual gait speed will be calculated based on a 10-meter walk distance. The investigators will provide individuals with a 14-meter path for walking to provide room for a "flying start." The participant will walk 14 meters, but gait speed will only be timed during the intermediate 10 meters. This will allow us to determine gait speed without the confounding factor of acceleration and deceleration.

SECONDARY OUTCOMES:
Feasibility- Recruitment | 12-weeks
  Acceptable recruitment will be assessed among those in the intervention. Acceptable recruitment is defined as 90% of targeted enrollment within 15 months of initiating recruitment efforts.
Physical Activity | 12-weeks
  Physical activity will be assessed as average steps per day, measured with a FitBit.
Acceptability- Usage Rating Profile-Intervention | 12-weeks
  Acceptability will be measured using the Usage Rating Profile-Intervention (URPI). A higher score indicates greater acceptability of the intervention. The URPI uses a 6-point Likert scale from 1 (strongly disagree) to 6 (strongly agree)
Muscular strength | 12-weeks
  Knee extension and plantar flexion strength will be assessed using a MicroFET 2 Hand-held Dynamometer
Perfusion | 12-weeks
  Cutaneous perfusion will be assessed on the dorsal and plantar surfaces of the foot using laser Doppler flowmetry using the PeriFlux System 5000
Glycemic control | 12-weeks
  Blood samples will be obtained by venipuncture of a vein in the upper extremity for HbA1c measurement.
Mobility | 12-weeks
  Community mobility will be assessed using the Life-Space Assessment (LSA).
Acceptability | 12-weeks
  Acceptability will be measured through a semi-structured interview.
Adherence to the exercise regimen | 12-weeks
  Adherence to the exercise regimen will be assessed using written logs of home-based exercise, attendance to virtual group exercise, and anonymized FitBit accounts.
Feasibility- Retention | 12-weeks
  Retention will be assessed among those in the intervention. Acceptable retention will be assessed by 80% participation in exercise intervention and study visits.
Community mobility | 12-weeks
  Community mobility will be assessed using the Life-Space Assessment (LSA).

CONTACTS AND LOCATIONS:
Overall Officials: Mary-Claire Roghmann, MD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Final data sets underlying all publications resulting from the proposed research will be shared outside VA. A limited dataset will be created and shared pursuant to a Data Use Agreement. Final data sets will be maintained locally until enterprise-level resources become available. Upon request, we will provide an electronic limited dataset to others in the scientific community with the implementation of appropriate data use agreements.
Supporting Information: Study Protocol, SAP
Time Frame: The protocol and SAP will be made available before analysis
Access Criteria: Implementation of appropriate data use agreements. Email the study PI, Dr. Mary-Claire Roghmann (mroghmann@som.umaryland.edu), to start the process.

REFERENCES:
- [Derived] Robinson GL, Drumheller J, Lydecker AD, Rammling B, Dennis EA, Addison O, Prior SJ, Beamer BA, Sorkin JD, Gottlieb HD, Trent K, Roghmann MC. Home-Based Exercise to Improve Functional Outcomes in Veterans With a Recently Healed Diabetic Foot Ulcer: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2025 Sep 23;14:e71237. doi: 10.2196/71237. PMID 40986852